CLINICAL TRIAL: NCT02231996
Title: Chronic Granulomatous Disease Study in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CGD-20140829
Record Dates: First submitted 2014-08-29; First posted 2014-09-04 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Granulomatous Disease, Chronic
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

GROUPS / COHORTS (1):
- gene mutation

SUMMARY:
CGD is a rare inherited primary immunodeficiency which is caused by the defect in one of the subunits of NADPH oxidase complex.We tend to collect and analyze Chinese CGD patients who are diagnosed in hospitals affiliated to Shanghai Jiao Tong University School of Medicine, including clinical feature, laboratory data and genetic information. we aim to find out clinical, distribution, genetic characteristic of CGD in Chinese population, etc., thus further improving the level of diagnosis and treatment for CGD.

ELIGIBILITY:
Inclusion Criteria:

* x-linked and AR-linked Chronic Granulomatous Disease
* history of life-threatening severe infections
* A functional assay demonstrating abnormal NADPH oxidase function or clinical history consistent with CGD

Exclusion Criteria:

* Presence of other primary immunodeficiency syndromes that do not meet the clinical and laboratory criteria for CGD.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: CGD patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
times of pneumonia | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai children's medical center, Shanghai, Shanghai Municipality, China